CLINICAL TRIAL: NCT01049594
Title: Evaluation of MR Imaging to Predict Neurodevelopmental Impairment in Preterm Infants
Brief Title: ePrime: Evaluation of Magnetic Resonance (MR) Imaging to Predict Neurodevelopmental Impairment in Preterm Infants
Acronym: ePrime
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: EudraCT 2009-011602-42; RP-PG-0707-10154 (Other Grant/Funding Number: The National Institute for Health Research)
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2010-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples containing DNA.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Preterm infants: Delivery at less than 33 completed weeks of gestation

SUMMARY:
Preterm infants face an uncertain future because premature birth often leads to problems with brain development and can cause cerebral palsy.

A trial needs to be done to see if Magnetic Resonance Imaging (MRI) helps families and professionals by predicting long term problems more accurately, allowing better targeting of care to children with problems and reassuring the parents of normal babies.

This programme will provide the evidence-base for the National Health System (NHS) policy on the use of magnetic resonance imaging of the brain for preterm infants.

DETAILED DESCRIPTION:
The trial will determine very accurately how well MRI predicts long-term problems, and it will assess whether it makes parents more or less anxious about their babies, and whether they seek more or less help in the first couple of years after birth,and see if the total cost to the NHS is increased by using MRI. It will also check up if there is a better way to do ultrasound examinations, and do a survey to see how much MRI is used in the United Kingdon (UK) and whether hospitals think they could provide it.

The core of the project is a study of preterm babies who will be referred to a specialist centre to have both ultrasound and MRI scans. Half the parents will be told the results of the MRI and half the parents the ultrasound. The programme will then ask them to fill in questionnaires or be interviewed about their stress levels and the amount of support they seek for their children until they are two years old, when the babies will be examined to see if MRI predicted their outcome accurately.

ELIGIBILITY:
Inclusion Criteria:

-Delivery at less than 33 completed weeks of gestation, estimated from early fetal ultrasonographic measurements as recommended in the National Institute of Clinical Excellence Guidelines: Antenatal Care for the Healthy Woman

Exclusion Criteria:

* Prior MR imaging
* Major Congenital Malformations
* Presence of Metallic Implants

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants delivered at less than 33 weeks of gestation. The North and South west London Perinatal Networks will provide a representative sample of the preterm infants cared for by the NHS.
Sampling Method: Non-Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2010-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
This programme will provide the evidence-base for NHS policy on the use of magnetic resonance (MR) imaging of the brain for preterm infants. | 5 years
  1. Determine with high precision the sensitivity and specificity of cerebral MR imaging for predicting neurodevelopmental impairment in the context of the NHS.
  2. Use a randomised design to compare the effect of MR and ultrasound imaging on total healthcare usage and costs, and assess its effect on unplanned and planned care.
  3. Compare the influence of MR- and ultrasound-based information on parental perceptions, stress and coping.
  4. Compare routine local bedside with specialist centralised ultrasound imaging.
  5. Survey current MR use and capacity in the NHS.
  6. Develop further novel MR methods to predict neurodevelopmental impairment.

CONTACTS AND LOCATIONS:
Overall Officials: David Edwards, Principal Investigator — Imperial College London
Locations (13):
- United Kingdom (13):
  - Croydon University Hospital, London
  - Barnet General Hospital, London
  - Northwick Park Hospital, London
  - Kingston Hospital NHS Trust, London
  - Guys & St Thomas NHS Trust Foundation, London
  - Epsom and St Helier University Hospital, London
  - St George's Healthcare NHS Trust, London
  - West Middlesex University Hospital, London
  - Ealing Hospital NHS Trust, London
  - Hillingdon Hopsital, London
  - Queen Charlotte's & Chelsea Hospital, London
  - St Marys Hospital, London
  - St. Peter's Hospital, Surrey

REFERENCES:
- [Derived] Edwards AD, Redshaw ME, Kennea N, Rivero-Arias O, Gonzales-Cinca N, Nongena P, Ederies M, Falconer S, Chew A, Omar O, Hardy P, Harvey ME, Eddama O, Hayward N, Wurie J, Azzopardi D, Rutherford MA, Counsell S; ePrime Investigators. Effect of MRI on preterm infants and their families: a randomised trial with nested diagnostic and economic evaluation. Arch Dis Child Fetal Neonatal Ed. 2018 Jan;103(1):F15-F21. doi: 10.1136/archdischild-2017-313102. Epub 2017 Oct 7. PMID 28988160
- [Derived] Harvey M, Nongena P, Edwards D, Redshaw M. 'We knew it was a totally at random thing': parents' experiences of being part of a neonatal trial. Trials. 2017 Aug 1;18(1):361. doi: 10.1186/s13063-017-2112-3. PMID 28764800